CLINICAL TRIAL: NCT05861765
Title: The Efficacy of Papaverine to Prevent Radial Artery Spasm During Transradial Cerebral Angiography: A Randomized Controlled Trial
Brief Title: The Efficacy of Papaverine to Prevent Radial Artery Spasm During Transradial Cerebral Angiography
Acronym: PASS
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 20230421
Record Dates: First submitted 2023-05-03; First posted 2023-05-17 (Actual); Last update posted 2023-06-12 (Actual); Status verified 2023-04

CONDITIONS: Radial Artery Spasm
Keywords: Radial artery spasm; Papaverine; Cerebral angiography
MeSH Terms: interventions — Papaverine; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Papaverine (Experimental): Slowly inject 10ml of papaverine hydrochloride solution (30mg/10ml) through the successfully implanted radial artery sheath, and continuously drip papaverine hydrochloride solution (60mg/500ml, 4ml/min) through the artery sheath during the operation. The compatible solutions are normal saline(0.9%);
  Interventions: Drug: Papaverine Hydrochloride
- Placebo (Placebo Comparator): After inserting the radial artery sheath, slowly inject 10ml normal saline(0.9%) through the artery sheath, and continuously drip normal saline(0.9%, 500ml, 4ml/min) through the artery sheath during the operation.
  Interventions: Drug: normal saline

INTERVENTIONS:
Drug: Papaverine Hydrochloride — Slowly inject 10ml of papaverine hydrochloride solution (30mg/10ml) through the successfully implanted radial artery sheath, and continuously drip papaverine hydrochloride solution (60mg/500ml, 4ml/min) through the artery sheath during the operation. The compatible solutions are normal saline(0.9%);
  Arms: Papaverine
Drug: normal saline — After inserting the radial artery sheath, slowly inject 10ml normal saline(0.9%) through the artery sheath, then continuously drip normal saline(0.9%, 500ml, 4ml/min) through the artery sheath during the operation.
  Arms: Placebo

SUMMARY:
Rationale:Papaverine is effective on radial artery spasm during transradial cerebral angiography.

Purpose: This multicenter, randomized, placebo-controlled, double blind, phase 2b trial aims to investigate the effect and safety of papaverine in treating radial artery spasm during transradial cerebral angiography.

DETAILED DESCRIPTION:
Radial artery spasm (RAS) is a common complication during transradial cerebral angiography. RAS can lead to severe pain and remains the most frequent cause of transradial angiography failure. There is currently no consensus on the prevention strategy for RAS.

Papaverine has anti vasospasm, sedative and analgesic effects. However, there is no evidence for the efficacy of papaverine in preventing RAS.

This multicenter, randomized, double blind, placebo-controlled trial aims to investigate the effect and safety of papaverine in treating radial artery spasm during transradial cerebral angiography.

ELIGIBILITY:
Inclusion Criteria:

1. All patients scheduled for cerebral angiography will be eligible for screening.
2. Participant is willing and is able to give informed consent for participating in the trial.
3. Male or Female, aged 18 years or above.

Exclusion Criteria:

1. Any patient with negative modified Allen test
2. Altered liver function
3. atrioventricular heart block III degree
4. Suspected or confirmed cerebral hemorrhage patients
5. Hemodynamic Instability : systolic pressure < 100 mmHg, heart rate > 100 bpm, tachycardia uncontrollable.
6. Patients with cerebral edema and increased intracranial pressure within 24 hours to 2 weeks after stroke
7. Coronary artery bypass grafting(CABG) operation history and whose right radial artery is missing as a "bridge vessel"
8. Severe skin musculoskeletal malformation of forearm or failure to complete radial artery puncture and sheath placement for other reasons
9. Hypersensitivity or contraindication to papaverine
10. Hypersensitivity or contraindication to nitroglycerine
11. Glaucomatous patients
12. Parkinson's disease patients
13. Women who are suspected or known to be pregnant or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2023-05-24 (Actual); Primary Completion 2023-09-30 (Estimated); Study Completion 2023-10-30 (Estimated)

PRIMARY OUTCOMES:
The incidence of RAS | Intraprocedural: From procedure start to application of radial band. Approximate time 30 to 90 minutes.
  The primary outcome of this trial is to evaluate the incidence of RAS during surgery. The operator assessed RAS on the basis of a questionnaire addressing the following five signs: persistent forearm pain, pain response on catheter manipulation, pain response to introducer withdrawal, difficult catheter manipulation after being "trapped" by the radial artery with considerable resistance on withdrawal of the introducer. RAS was considered to be indicated by the presence of at least 2 of these 5 signs or by the presence of just 1 when the operator considered it necessary to administer other spasmolytic agent.

SECONDARY OUTCOMES:
The pain intensity of the right forearm | Intraprocedural: From procedure start to application of radial band. Approximate time 30 to 90 minutes.
  Evaluate the pain intensity of the right forearm during the surgery based on the Numerical Rate Scale(NRS), which evaluates the worst pain during the surgery from "0" indicating "No Pain" to "10" indicating "Pain as bad as you can imagine".
The incidence of transradial approach failure | Intraprocedural: From procedure start to application of radial band. Approximate time 30 to 90 minutes.
  Transradial approach failure is defined as needing to change the route to complete the surgery.

OTHER OUTCOMES:
The risk of death, non fatal myocardial infarction, and stroke | Within 1 week after surgery
  The incidence of death, non fatal myocardial infarction, and stroke
Severe systemic hypotension | Within 24 hours after surgery or during surgery
  Systolic blood pressure decrease>30 mmHg or need to use vasopressor medication
Complications at the puncture site | Within 24 hours after surgery
  The incidence of complications at the puncture site

CONTACTS AND LOCATIONS:
Overall Officials: Yamei Tang, PhD, Study Chair — Department of Neurology, Sun Yat-sen Memorial Hospital, Sun Yat-sen University
Locations (1):
- Sun Yat-sen Memorial Hospital, Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Pan D, Yang J, Liu M, Xu Y, Feng J, Li H, Luo W, He B, Xiao S, Yang X, Tang Y. Efficacy of Papaverine to Prevent Radial Artery Spasm During Transradial Cerebral Angiography (PASS): rationale and design. Stroke Vasc Neurol. 2025 Sep 10:svn-2024-003659. doi: 10.1136/svn-2024-003659. Online ahead of print. PMID 40930776